CLINICAL TRIAL: NCT03726593
Title: Multicenter Therapeutic Efficacy Assessment of Pyronaridine-Artesunate (Pyramax®) and New Drug Combinations With Atovaquone-Proguanil for the Treatment of Uncomplicated P. Falciparum Malaria in Cambodia
Brief Title: Drug Combinations of Atovaquone-Proguanil (AP) With ACT
Acronym: APACT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Collaborators: National Center for Parasitology, Entomology, and Malaria Control (CNM) (Unknown); Naval Medical Research Unit-2 (NAMRU-2) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WR2530
Record Dates: First submitted 2018-10-16; First posted 2018-10-31 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Plasmodium Falciparum Malaria (Drug Resistant)
Keywords: malaria; plasmodium falciparum; malarone; atovaquone; mefloquine; pyramax; pyronaridine; combination treatment; triple therapy; multidrug resistant malaria
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination; atovaquone, proguanil drug combination

STUDY DESIGN:
Intervention Model Description: Randomized, open-label clinical trial to evaluate the tolerability and clinical and parasitological responses after treatment of Pf and/or mixed infections (Pf/Pv) in volunteers with uncomplicated malaria. The assignment of volunteers will be 1:1:1 for ASPY (Pyramax), AP+ASPY (AP+Pyramax), and AP+ASMQ. All study drug administration will be by directly observed therapy (DOT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASPY (Experimental): Artesunate-pyronaridine, once daily for three days, following standard weight-based dosing per drug label. All volunteers with P.f monoinfection will receive single dose of primaquine (PQ) (15 mg) for transmission blocking.
  Interventions: Drug: Artesunate and Pyronaridine
- AP+ASPY (Experimental): Atovaquone-Proguanil (AP) + Artesunate-Pyronaridine (ASPY), once daily for three days, following standard weight-based dosing per drug label for each drug. All volunteers with P.f monoinfection receive single dose of PQ (15 mg) for transmission blocking
  Interventions: Drug: Atovaquone Proguanil and Artesunate Pyronaridine
- AP+ASMQ (Experimental): Atovaquone-Proguanil (AP) + Artesunate-Mefloquine (ASMQ); ASMQ once daily for three days (D0, D1, D2), following standard weight-based dosing per drug label. Subsequently, volunteers continue their treatment with AP once daily starting on day 3, for three additional days (D3, 4, 5). All volunteers with P.f monoinfection receive single dose of PQ (15 mg) for transmission blocking.
  Interventions: Drug: Atovaquone Proguanil and Artesunate Mefloquine

INTERVENTIONS:
Drug: Artesunate and Pyronaridine — Standard weight based dosing
  Arms: ASPY
Drug: Atovaquone Proguanil and Artesunate Pyronaridine — Both drugs (AP) and (ASPY) are administered once a day, on days 0, 1, and 2.
  Arms: AP+ASPY
Drug: Atovaquone Proguanil and Artesunate Mefloquine — Sequential treatment with ASMQ (on days 0, 1, and 2) followed by the treatment with AP for 3 more days (total 6 days treatment)
  Arms: AP+ASMQ

SUMMARY:
Investigators are conducting this study due to recent reports of many of existing malaria drugs becoming less effective for treatment of malaria. The drugs may not always kill all the parasites, therefore not all patients with malaria are being cured. The main objective of the study is to find out which malaria drugs and what drug combinations are still effective in Cambodia, an area of multi-drug resistance where 4-5 artemisinin-based combination therapies have shown inadequate response, below that established by the World Health Organization (WHO). New drug combinations (taking more than one drug for malaria at the same time), as long as well tolerated, can provide cure in patients that harbor parasites not responsive to standard first-line medications. Human genetic testing will be done to identify patients who may have suboptimal response to treatments and to study the differences in human gene expression to explain why some persons are at higher risk of complications during treatment. Markers of drug resistance to commonly used antimalarial drugs will also be evaluated and shared with national malaria program (CNM) to better guide future malaria treatment decisions in Cambodia.

DETAILED DESCRIPTION:
Efficacy to drugs that are currently available and new antimalarial candidates that are in development are threatened by multidrug resistant (MDR) malaria parasites, widely prevalent in Cambodia. Without effective interventions, MDR malaria can pose a substantial public health threat in the years to come. Therefore, accurate, timely and relevant data on antimalarial drug resistance is of critical importance. Prompt, effective and well-tolerated treatment remains one of the cornerstones in the malaria case management. Recent malaria outbreak in Thailand and rise of malaria cases observed in Cambodia in 2017 has brought to the forefront the urgency with which new drug candidates and new combination drug treatments must be identified; otherwise, patients may be left with ineffective treatments. Lack of available alternatives has a potential to result in significant setback to the recent gains in malaria control and malaria elimination efforts. Innovative approaches to treatment proposed here, using current ACTs in combination with non-ACT drugs, such as atovaquone-proguanil, need to be investigated to assess drug tolerability and overall efficacy when used under combination treatment. By early investment in the studies of drugs such as pyronaridine-artesunate (ASPY), in combination with other antimalarials, and drug combinations proposed under this protocol, this study will try to provide the latest evidence on the interventions that are most likely to work, even in areas of MDR, such as Cambodia, and along the Cambodia-Thai border. It is hoped that our approach for using combination treatments will not only provide more effective treatments, but it might prolong the lifespan of the remaining antimalarials and delay the spread of MDR malaria to neighboring countries.

ELIGIBILITY:
Inclusion Criteria:

* Understands Khmer spoken language
* Male or female (18 to 70 years old)
* Microscopic confirmation of asexual stages of Pf or mixed infection with Pf, with baseline asexual parasite densities between 100/µL to 200,000/µL
* Able to take oral medications
* Hemoglobin on day of enrollment ≥9.0 g/dL
* Agree to follow-up for the anticipated study duration, including a minimum of 3 nights at the medical treatment facility (inpatient hospitalization) and weekly follow-up visits for at least 6 weeks
* If the volunteer is on active duty in the military, the volunteer has written permission from their supervisor or states to have been authorized by his/her supervisor or the local commander to participate; and allow study staff to contact their supervisor to confirm this information

Exclusion Criteria:

* Known allergic reaction to any of the study drugs or history of severe intolerance to any of the antimalarials used in this study.
* Pregnant or lactating females and females of childbearing potential who do not agree to use an acceptable form of contraception during the study period and for 6 weeks following the last dose of the study drug.
* Symptoms of severe vomiting (inability to tolerate oral fluids or oral medications during the previous 8 hours or vomiting >3 times in the last 24 hrs).
* Diagnosis of severe malaria
* Abnormal liver function tests i.e AST or ALT or total bilirubin > 1.5 upper limit of normal (ULN) with nausea AND right upper quadrant abdominal pain OR jaundice on exam
* Isolated AST or ALT or Total Bilirubin >2x ULN
* Known significant cardiovascular, liver or renal abnormality or any other clinically significant illness, which in the opinion of the investigator would place the volunteer at significantly higher risk
* Treatment for malaria within the last 4 weeks
* Unable to provide informed consent
* Judged by the investigator to be otherwise unsuitable for study participation (to include, but not limited to, taking other medications that are known to cause serious drug-drug interactions with the study drugs, as determined by the study physician, or having suspected medical condition or taking other drugs that may affect test results interpretation or put the volunteer at much higher risk)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
42-day polymerase chain reaction (PCR) corrected adequate clinical and parasitological response (ACPR), following treatment with ASPY and new drug combinations (AP+ACTs). | 6 weeks

SECONDARY OUTCOMES:
Prevalence of molecular markers of drug resistance | Day of enrollment and day of malaria recurrence up to 8 weeks
Drug susceptibility testing of parasite isolates against standard antimalarial drugs | Day of enrollment and day of malaria recurrence up to 8 weeks
  Ex vivo drug susceptibility testing
Pharmakokinetics of each study drug - (Cmax) | multiple time points up to 8 weeks
  Peak plasma concentration (Cmax) for study drugs
Pharmakokinetics of each study drug - (AUC) | multiple time points up to 8 weeks
  Area under the plasma concentration versus time curve (AUC)
Pharmakokinetics of each study drug - volume of distribution | multiple time points throughout 6 weeks of follow up
  volume of distribution for study drugs
Pharmakokinetics of each study drug - (T1/2) | multiple time points up to 8 weeks
  elimination half-life (T1/2) for study drugs
Kaplan Meier survival analysis of asexual blood stage parasitemia and sexual stage gametocytes | 6 weeks
Gametocyte carriage rates on days 0, 1, 2, 3, and weeks 1 through 6 for each treatment arm | Days 0, 1, 2, 3, and weekly, up to week 8
The incidence of hepatotoxicity events for each treatment arm | Day 3 and week 6
  Alanine aminotransferase (ALT)>5 times the upper limit of normal (ULN) or percent of volunteers meeting the Hy's law definition (ALT or aspartate aminotransferase [AST] >3 x ULN and total bilirubin >2 x ULN) at any post-dose time point within 6 weeks of follow up
Rates of treatment-related adverse events | 6 weeks
Severity of treatment-related adverse events | 6 weeks
  Grade 1 - mild, Grade 2 - moderate, Grade 3 - severe, Grade 4- life threatening
Number of participants who say they are willing to take the same drug combination in the future | day 2 and week 6
Point efficacy with 95% Confidence Interval against blood stage malaria infection classified according to the WHO malaria treatment outcome classifications (ETF, LTF, LCTF, LPTF) | 4 weeks, 6 weeks, and 8 weeks
Incidence of Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency | Enrollment
  Comparative incidence of G6PD deficiency in the study population as determined by G6PD rapid-diagnostic tests (RDTs) and quantitative tests, to include sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV) for each of the point-of-care tests against 10%, 30%, and 60% thresholds of normal G6PD activity
Number of infected mosquitos following membrane feeding | Day 0, Day 3, Day 7, and on day of malaria recurrence up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Wojnarski, MD, Principal Investigator — Armed Forces Research Institute of Medical Sciences (AFRIMS) Bangkok, Thailand
Locations (3):
- Cambodia (3):
  - Anlong Veng Referral Hospital, Anlong Veaeng
  - Kratie Referral Hospital, Kratié
  - Stung Treng Referral Hospital, Stung Treng

IPD SHARING:
Plan to Share IPD: No
The study site will maintain appropriate medical and research records for this trial until completion of the study, in compliance with Section 4.9 of International Conference on Harmonization E6 Good Clinical Practices, and institutional requirements. The investigators and other study personnel assigned from National Center for Parasitology, Entomology and Malaria Control (CNM), Armed Forces Research Institute of Medical Sciences (AFRIMS) and Naval Medical Research Center NMRC-Asia and their respective representatives are authorized access to the study data as part of their duties. The database may be shared with other collaborators, on a mutually agreed basis. Sharing and publication of the data with other parties can be done only after inter-institutional agreements are in place. The research findings may be disseminated to policy makers and other researchers for an informed decision on drug policy for the treatment of malaria.